CLINICAL TRIAL: NCT02725060
Title: Autoimmune Basis for Postural Tachycardia Syndrome
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: University of Oklahoma (Other)
Responsible Party: Principal Investigator, Luis E Okamoto, Research Instructor, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 151791
Record Dates: First submitted 2016-02-22; First posted 2016-03-31 (Estimated); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Postural Orthostatic Tachycardia Syndrome; Postural Tachycardia Syndrome; Tachycardia; Arrhythmias, Cardiac; Autonomic Nervous System Diseases; Orthostatic Intolerance; Cardiovascular Diseases; Primary Dysautonomias
Keywords: POTS; Orthostatic Intolerance; Orthostatic Tachycardia
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Tachycardia; Arrhythmias, Cardiac; Autonomic Nervous System Diseases; Orthostatic Intolerance; Cardiovascular Diseases; Primary Dysautonomias | interventions — Phenylephrine; Isoproterenol; Blood Specimen Collection; Blood Pressure Monitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autonomic and Antibody Assessments (Experimental): On up to 3 study days, POTS patients and control subjects will have several tests to assess autonomic function and to detect the presence of autoantibodies to adrenergic receptors. The following tests will de done but in some participants it may not be necessary to do all of them. The investigator will discuss with each participant which particular tests will be done in each particular case:
  * Posture study with blood samples for autoantibody testing
  * 24-hour heart rhythm and blood pressure monitoring
  * autonomic function tests
  * Quantitative Axonal Sudomotor Reflex Testing
  * Total blood volume assessment
  * Pharmacologic testing with phenylephrine
  * Pharmacologic testing with isoproterenol
  * Cardiac output with rebreathing
  * Assessment of splanchnic capacitance
  * Microneurography
  Interventions: Drug: phenylephrine; Drug: isoproterenol; Radiation: 25 micro-Ci of radiation; Procedure: Posture study with blood samples; Procedure: 24-hour heart rhythm and blood pressure monitoring; Procedure: Quantitative Axonal Sudomotor Reflex Testing; Procedure: Autonomic function tests; Other: Rebreathing test; Other: Assessment of splanchnic capacitance; Procedure: microneurography

INTERVENTIONS:
Drug: phenylephrine — Phenylephrine is a selective α1-adrenergic receptor agonist. It will be given in IV bolus injections starting from 12.5 ug. Incremental doses will be given every ~3 min up to 800 ug or until systolic blood pressure increases by 25 mmHg
Drug: isoproterenol — Isoproterenol is non-selective beta-adrenergic agonist. It will be given in IV bolus injections starting from 0.025 ug. Incremental doses will be given every ~3 min until heart rate increases by 25 bpm. This intervention is optional.
  Other Names: isuprel; isoprenaline
Radiation: 25 micro-Ci of radiation — Using injection of iodinated I-131 tagged human serum albumin nominally 25 micro-Ci of radiation, blood samples are drawn before and 30 minutes after injection.
  Other Names: DAXOR
Procedure: Posture study with blood samples — Blood pressure and heart rate will be measured while supine and then while standing for up to 30 minutes. Blood will be drawn in each position to measure hormones that regulate blood pressure and blood volume. An additional sample will be collected in the supine position for the autoantibody assessment.
  Other Names: orthostatic challenge; orthostatic stress test
Procedure: 24-hour heart rhythm and blood pressure monitoring — Blood pressure, heart rate and ECG monitoring for 24 hours
  Other Names: 24 Holter
Procedure: Quantitative Axonal Sudomotor Reflex Testing — The QSART assesses the ability of sympathetic nerve terminals in the skin to release acetylcholine and increase sweat production. The test is performed at 4 sites over the forearm, proximal lateral leg, medial distal leg and proximal foot.
  Other Names: QSART; sweat test
Procedure: Autonomic function tests — The autonomic function tests will determine how well the autonomic nervous system regulates blood pressure and heart rate. These tests include breathing deeply for two minutes, breathing fast for 30 seconds, maintaining a handgrip for 3 minutes, breathing against pressure for 15 seconds, and placing the hand in ice water for 1 minute. In addition, participants will be tilted up on a tilt table for up to 10 minutes while recording their heart rate, blood pressure and cardiac output.
Other: Rebreathing test — Cardiac output will be measured using the rebreathing technique (Innocor)
  Other Names: cardiac output measurement
Other: Assessment of splanchnic capacitance — Splanchnic capacitance will be assessed using cpap and body impedance to construct pressure volume curves
Procedure: microneurography — microneurography will be measured in the peroneal nerve to assess sympathetic activity.
  Other Names: msna

SUMMARY:
The purpose of this study is to see if some people with postural tachycardia syndrome (POTS) have higher levels of immune proteins (autoantibodies) directed against receptors of the autonomic nervous system, and if these autoantibodies make a difference in their POTS symptoms. The investigators also want to see if the levels of these autoantibodies stay the same over time.

DETAILED DESCRIPTION:
Postural tachycardia syndrome (POTS) is a debilitating disorder resulting from cardiovascular autonomic dysfunction, has many causes and is very difficult to treat effectively. The investigators have identified the presence of autoantibodies (immune proteins) directed against some receptors of the autonomic nervous system that can cause patient's symptoms on standing.

The present study is designed to test the hypothesis that patients with POTS harbor functional autoantibodies to adrenergic receptors that lead to an excessive tachycardia characteristic of POTS. For this purpose, this study will define the prevalence, burden, and the in vivo physiological significance of these adrenergic antibodies in a well-phenotyped and representative cohort of patients with POTS and a matched cohort of healthy control subjects, and will characterize the stability of these autoantibodies over time in affected POTS patients.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years old
* Postural Tachycardia Syndrome: Heart rate increase >30 bpm from supine within 10 min of standing, in the absence of orthostatic hypotension (>20/10 mmHg fall in blood pressure), with chronic symptoms (> 6 months), and in the absence of other acute cause of orthostatic tachycardia.
* Able and willing to provide informed consent
* Female premenopausal subjects must utilize adequate birth control and willingness to undergo serum beta-hCG testing
* The subject must understand and be able to comply with the study procedures and restrictions.

Exclusion Criteria:

* Hypertension (>150 mmHg systolic and >100 mmHg diastolic) based on history or findings at screening.
* Orthostatic hypotension (consistent drop in blood pressure >20/10 mmHg with 10 min stand)
* Pregnancy
* Cardiovascular disease, such as myocardial infarction within 6 months, angina pectoris, significant arrhythmia (sinus tachycardia is not excluded), deep vein thrombosis, pulmonary embolism
* History of serious neurologic disease
* History or presence of significant immunological or hematological disorders
* Clinically significant gastrointestinal impairment that could interfere with dietary compliance or drug absorption
* Impaired hepatic function (aspartate amino transaminase and/or alanine amino transaminase >1.5 x upper limit of normal range)
* Impaired renal function (serum creatinine >1.5 mg/dL)
* Hematocrit <28%
* Current or concurrent disease that could affect the absorption, action or disposition of the drug, or clinical or laboratory assessments.
* Any underlying or acute disease requiring regular medication that could possibly pose a threat to the subject or make implementation of the protocol or interpretation of the study results difficult
* Inability to comply with the protocol

Healthy control subjects will be healthy, non-smoking and on no chronic medications at the time of the study. Healthy control subjects will be group-matched to the POTS patients for age and gender. We will attempt to study female patients in the first half of their menstrual cycle to minimize cyclical variability.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Autoantibody levels | up to 10 minutes
  Blood samples collected while supine during the posture study will be analyzed for autoantibody positivity in POTS patients and control subjects.
Blood pressure after phenylephrine boluses | 1-2 minutes after bolus injections
Heart rate after isoproterenol boluses | 1-2 minutes after bolus injections
Orthostatic change in heart rate | up to 10 minutes
  Difference between standing and supine heart rates.

SECONDARY OUTCOMES:
Blood pressure response during phase IV of the Valsalva maneuver | up to 10 minutes
Hear rate response during phase IV of the Valsalva maneuver | up to 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Luis Okamoto, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (2):
- United States (2):
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Autonomic Dysfunction Center, Nashville, Tennessee